CLINICAL TRIAL: NCT06582251
Title: The Effects of High-Intensity Functional Training Versus Traditional Strength Training or Concurrent Training on Performance and Readiness in Tactical Populations
Brief Title: The Effects of High-Intensity Functional Training in Tactical Populations
Acronym: HIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Strength and Conditioning Association (Other)
Responsible Party: Principal Investigator, Shawn M. Arent, Professor and Chair of Exercise Science Department, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00137947
Record Dates: First submitted 2024-08-27; First posted 2024-09-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy
Keywords: high-intensity functional training; tactical; military

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Functional Training (Experimental): Training will include power and strength movements, then 30 minutes of metabolic conditioning training comprised of whole-body multi-joint movements.
  Interventions: Behavioral: High-intensity functional training
- Traditional Resistance Training (Active Comparator): This group will perform traditional resistance training.
  Interventions: Behavioral: Traditional resistance training
- Concurrent Training (Active Comparator): This group will perform traditional resistance training followed by 20 minutes of running, high intensity intervals.
  Interventions: Behavioral: Concurrent training

INTERVENTIONS:
Behavioral: High-intensity functional training — Participants assigned to this group will undergo 8 weeks of high-intensity functional training.
  Arms: High Intensity Functional Training
Behavioral: Traditional resistance training — Participants assigned to this group will undergo 8 weeks of traditional strength and hypertrophy training.
  Arms: Traditional Resistance Training
Behavioral: Concurrent training — Participants assigned to this group will undergo 8 weeks of traditional strength and hypertrophy training followed by high-intensity interval aerobic training.
  Arms: Concurrent Training

SUMMARY:
The purpose of this study is to investigate the effects of high-intensity functional training (HIFT) as compared to traditional resistance training (RT) and concurrent training consisting of RT and high-intensity interval training (HIIT) on physical performance metrics, body composition, and mental and physical readiness of tactical personnel.

DETAILED DESCRIPTION:
This study assesses the impact of 8-weeks of high-intensity functional training (HIFT) as compared to traditional resistance training (RT) and concurrent training consisting of RT and high-intensity interval training (HIIT) on various performance outcomes. The main questions the study aims to answer are:

* Evaluate the distinct effects of HIFT, RT, and RT plus HIIT over eight weeks on physical performance and body composition measures in tactical men and women.
* Determine the distress, training load, and physical readiness associated with each of the three distinct training interventions over eight weeks.

Participants will:

* Take part in 10-weeks total of study-related activity.
* Complete four total sessions of pre and post-testing sessions, which include body composition, maximal oxygen uptake testing (VO2max), upper and lower body maximal strength, and lower body power.
* Be randomly assigned to an exercise training intervention.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 35 (inclusive) and enrolled in a reserve officer training corps program.
* Subject has provided written and dated informed consent to participate in the study.
* Subject is in good health as determined by medical history and is cleared for exercise.
* BMI between 17.0 and 29.9 kg/m2.
* "Good" category or greater for their aerobic capacity according to the American College of Sports Medicine (ACSM) normative data for their age and sex as measured at their baseline visit.

Exclusion Criteria:

* Participants with any musculoskeletal injuries that would prevent completion of these exercise programs.
* Participants with any metabolic disorder, including known electrolyte abnormalities, uncontrolled diabetes, uncontrolled thyroid disease, adrenal disease, or hypogonadism.
* Participants with a history of hepatorenal, musculoskeletal, autoimmune, or neurologic disease.
* Participants who have lost or gained greater than eight pounds within three months prior to study enrollment.
* Participants currently taking hyperlipidemic, hypoglycemic, anti-hypertensive, or anti-coagulant medications.
* Participants who are pregnant or lactating.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in body composition body fat percentage. | Baseline and Week 10
  Body fat percentage via air-displacement
Changes in body composition fat-free mass. | Baseline and Week 10
  Fat-free mass via air-displacement plethysmography.
Changes in body composition dry fat-free mass. | Baseline and Week 10
  Dry fat-free mass via air-displacement plethysmography and bio-electrical impedance.
Changes in upper body strength. | Baseline and week 10
  Upper body strength assessed by 1 repetition maximum bench press.
Changes in lower body strength. | Baseline and week 10
  Lower body strength assessed by isometric mid-thigh pulls on bilateral force plates.
Changes in maximal oxygen consumption. | Baseline and week 10
  Changes in VO2max measured by maximal graded exercise test with indirect calorimetry.
Changes in ventilatory threshold. | Baseline and week 10
  Changes in ventilatory threshold measured by maximal graded exercise test with indirect calorimetry.
Changes in velocity at VO2 max. | Baseline and week 10
  Assessed by maximal graded exercise test with indirect calorimetry.

SECONDARY OUTCOMES:
Internal training load between groups. | Every training session over the 8-week intervention period will be included in this calculation.
  Assessed by heart rate chest strap using Edwards training impulse calculation.
Changes in training distress | Baseline, once per week for the 8 training weeks.
  Overall training distress and subscales including depressed moods, vigor, physical signs and symptoms, sleep disturbances, perceived stress, and general fatigue using the multicomponent training distress scale, scaled 0 - 110 with higher scores indicating more distress.
Changes in anaerobic power. | Baseline, once per week for the 8 training weeks.
  Measured by countermovement jump through bilateral force plates.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina Sport Science Lab, Columbia, South Carolina, United States